CLINICAL TRIAL: NCT03265106
Title: A Clinical Study Evaluating the Safety and Efficacy of BinD19 Treatment in Relapse or Refractory Childhood Acute Lymphoblastic Leukemia and Lymphoma Subjects
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of BinD19 Treatment in Childhood R/R ALL and Lymphoma Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen BinDeBio Ltd. (Industry)
Collaborators: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017FDEK-BinD19
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Relapsed B-cell Acute Lymphoblastic Leukemia, Childhood; Refractory B-cell Acute Lymphoblastic Leukemia, Childhood; Relapsed/Refractory B-cell Lymphoma, Childhood
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BinD19 (Experimental): BinD19 (autologous T cells transduced with CD19 TCR-ζ/4-1BB vector) administered as an IV infusion on days 0, 1 and 2 in the absence of disease progression or unacceptable toxicity. Minimum/ maximum dose: 1x10^6/kg / 1x10^7/kg administered to childhood patients with R/R B cell Acute Lymphoblastic Leukemia (ALL) or Lymphoma.
  Interventions: Biological: BinD19

INTERVENTIONS:
Biological: BinD19 — Autologous T cells purified from the peripheral blood mononuclear cells of subjects, transduced with TCR- ζ/4-1BB lentiviral vector, expanded in vitro and then frozen for future administration.

SUMMARY:
This is a single arm, open-label, uni-center, phase I/II study to determine the safety and efficacy of an experimental therapy called BinD19 cells in childhood patients with B-cell acute lymphoblastic leukemia or lymphoma, who are chemo-refractory, relapsed after allogeneic SCT, or are otherwise ineligible for allogeneic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD19+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.
* CD19+ leukemia or lymphoma
* Not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor
* Follicular lymphoma, previously identified as CD19+:
* Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc)
* ECOG result is 0, 1 or 2.
* With normal heart, liver and kidney functions.
* Negative serum DNA for EBV and CMV; negative antigen for HBV; negative serum antibody for HCV, HIV and syphilis.
* Negative in pregnancy test (female subject only).

Exclusion Criteria:

* ECOG result is 3, 4 or 5.
* Pregnant or lactating female
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* HIV infection
* Enrolled to other clinical study in the last 4 weeks.
* Subjects with systemic auto-immune disease or immunodeficiency.
* Subjects with CNS diseases.
* Subjects with secondary tumors.
* Subjects with tumor infiltration in liver, brain or GI tract.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events [Safety and Feasibility] | Study treatment until Week 24
  To evaluate the safety and feasibility of BinD19 CAR-T cells in patients with refractory /relapsed B-cell acute lymphoblastic leukemia or lymphoma.

SECONDARY OUTCOMES:
Overall Response [Efficacy] | 5 years
  Efficacy assessments for ALL were performed based on bone marrow and blood morphologic criteria and physical examination findings. Efficacy assessments for Lymphoma were based on tumor load, B cell number and immunoglobulins.

CONTACTS AND LOCATIONS:
Overall Officials: ZHONG HUA YANG, Study Director — Shenzhen BinDeBio Ltd.
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No